CLINICAL TRIAL: NCT06421766
Title: Retrospective Study of Outcomes With 3 mm Implant for Percutaneous Bone-anchored Hearing System (BAHS) Procedures
Brief Title: Retrospective Study of Outcomes With 3 mm Implant for Percutaneous BAHS Procedures
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC122
Record Dates: First submitted 2024-04-23; First posted 2024-05-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- 3mm implant: Patients recieving a 3mm long implant
  Interventions: Device: BAHS
- 4mm implant: Patients recieving a 4mm long implant
  Interventions: Device: BAHS

INTERVENTIONS:
Device: BAHS — Implantation of a percutaneous bone-anchored hearing system

SUMMARY:
This retrospective study is conducted to gain more knowledge on use and complications of 3mm long implants used in percutaneous (through the skin) bone-anchored hearing system (BAHS) surgeries in adults. Patients included have already been treated and recieved an implant with the wide diameter (Ø: 4.5 mm) design, either of 3- or 4mm length. The main purpose of the study is to investigate implant survival three months after implantation.

DETAILED DESCRIPTION:
BAHS systems are intended for patients with conductive or mixed hearing loss, and for patients with single-sided deafness. In BAHS surgery, an implant - coupled to a skin-penetrating abutment - is implanted in the bone behind the ear and is later loaded with a sound processor. The sound processor transforms sound waves to sound vibrations that are transferred through the skull bone to the inner ear(s)/cochlea. Thus, sound can be transmitted directly to the cochlea and bypass any problems in the ear canal or middle ear. Today, more than 400,000 implantations have been made around the world and the long-term success rate of BAHS surgery is high, with a low rate of major complications.

Over the years, both implant design and surgical techniques have developed, with improved patient outcomes as a result. Wider diameter implants, 4.5mm in diameter, increased the implant stability and have become standard. The implants exist in two different lengths, 3- and 4mm, to accomodate for different bone thickness. The shorter implant has primarily been used for (young) children and for adults with thinner bone. The aim of this restrospective study is to investigate the outcomes after implantation of a 3mm implant in an adult population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥19 years) receiving percutaneous BAHS treatment using an implant with the wide diameter (Ø: 4.5 mm) design.

Exclusion Criteria:

* Patient undergoing re-implantation due to previous failure of osseointegration or other spontaneous implant loss.
* Patient undergoing conversions from passive transcutaneous devices (i.e. BAHA Attract) to active percutaneous devices (using an abutment), using the same implant for attachment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have already obtained surgical intervention with a percutaneous bone anchored hearing system.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Implant survival | 3 months after implant surgery
  Implant in place in skull bone at 3 months (Yes/No).

SECONDARY OUTCOMES:
Implant survival | Through study completion, with minimum 3 months
  Implant in place in skull bone at end of observation (Yes/No).
Number and type of intraoperative events | During surgery
  Assessment of intraoperative events during surgery by the investigator. Will be presented in a frequency table.
Number and type of postoperative events | Up to 3 months
  Assessment of postoperative events during the initial postoperative period (0-3 months) by the investigator. Will be presented in a frequency table.
Time to sound processor loading | Up to 3 months
  Time from surgery to sound processor loading

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G Pappas, MD, Principal Investigator — Alabama Ear Specialists
Locations (1):
- Alabama Ear Specialists, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No